CLINICAL TRIAL: NCT00249782
Title: A Phase II, Randomized, Partial-Blind, Parallel-Group, Active- and Vehicle-Controlled, Multicenter Study of the Safety and Efficacy of ACZONE™ (Dapsone) Gel, 5% in Subjects With Papulopustular Rosacea
Brief Title: A Phase II, Randomized Study of ACZONE™ (Dapsone) Gel, 5% for Papulopustular Rosacea.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACZ ROS 01
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Rosacea
Keywords: rosacea, Papulopustular Rosacea,erythema, dapsone
MeSH Terms: conditions — Rosacea; Erythema | interventions — Dapsone; Gels; Metronidazole

INTERVENTIONS:
Drug: Vehicle control, 2x/day
Drug: ACZONE (dapsone) Gel, 5%, 2x/day
Drug: ACZONE (dapsone) Gel, 5%, 1x/day
Drug: MetroGel® (metronidazole gel), 1.0% 1x/day
Drug: ACZONE (dapsone) Gel, 5%, 1x/day (AM) + MetroGel (metronidazole gel), 1.0%, 1x/day (PM)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of ACZONE™ gel compared to placebo (inactive substance), MetroGel® and a combination of ACZONE™ gel and MetroGel® for the treatment of rosacea.

ACZONE™ gel, 5% is a topical (applied to the skin) medication that is approved by the United States Food and Drug Administration (FDA) for the treatment of acne vulgaris in people 12 years and older. The use of ACZONE™ for the treatment of rosacea is investigational. An investigational use is one that is not approved by the FDA.

Subjects will apply the study treatment for 12 weeks. Efficacy assessments will be performed at baseline and Weeks 2, 4, 8, and 12. Laboratory assessments will be conducted at baseline and Week, 2, 4 and 12.

DETAILED DESCRIPTION:
Study Objective:

•To evaluate the safety and preliminary efficacy of ACZONE in subjects with papulopustular rosacea

Study Population: Approximately 400 male and female subjects will be enrolled at 27 study centers in the United States.

Study Treatment: Subjects will be randomized to 1 of 5 treatment regimens. Subjects will receive study medication for 12 weeks. Study participation is 13 weeks (5 clinic visits and 1 telephone follow-up).

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, subjects must fulfill all of the following criteria:

1. Men or women ≥18 years of age.
2. A diagnosis of papulopustular rosacea, with ≥10 inflammatory lesions (papules and/or pustules) above the mandibular line at baseline.
3. An Investigator Global Assessment (IGA) score ≥2
4. In good physical and mental health.
5. Signature of an approved informed consent form for the study and HIPAA authorization (if applicable).
6. Willingness to comply with the protocol.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. A skin examination reveals the presence of another skin disease and/or condition (excessive facial hair, excessive scarring, sunburn, or other disfigurement) located on the face that would confound the evaluation of the rosacea condition.
2. Current or past ocular rosacea, such as conjunctivitis, iritis, and keratitis, of sufficient severity to require topical or systemic antibiotics.
3. Treatment with topical antibiotics, topical steroids and other topical rosacea treatments on the face within 14 days of Baseline and throughout the study.
4. Treatment with systemic steroids within 30 days of Baseline and throughout the study.
5. Treatment with any systemic antibiotics within 30 days of Baseline and throughout the study.
6. Treatment with any systemic medication or therapy known to affect inflammatory responses within the 30 days prior to Baseline or throughout the study.
7. Treatment with topical retinoids within 30 days or systemic retinoids within 180 days of Baseline and throughout the study.
8. Treatment with physical modalities that could benefit rosacea are prohibited within 30 days of Baseline and throughout the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2005-11; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Efficacy: Percent change and change from baseline in inflammatory lesion counts;
"Success" rate, defined as proportion of subjects with a score of 0 or 1 and at least a 2 point improvement from baseline on the IGA scale;
Erythema & telangiectasia scores;
Lesion counts over time

SECONDARY OUTCOMES:
Safety: Adverse events and concomitant medications; Local symptom scores; Hematology and chemistry laboratory parameters; Vital signs
Other: Plasma dapsone concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Steven Garrett, MS, DDS, Study Director — QLT USA, Inc.
Locations (26):
- United States (26):
  - Radiant Research, Birmingham, Alabama
  - Radiant Research, Tucson, Arizona
  - East Bay Dermatology Medical Group, Inc., Fremont, California
  - Therapeutics Clinical Research, San Diego, California
  - Clincial Research Specialists, Inc., Santa Monica, California
  - Cherry Creek Research, Inc, Denver, Colorado
  - The Savin Center, PC, New Haven, Connecticut
  - Visions Clinical Research, Boynton Beach, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - FXM Research, Miami, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Welborn Clinic, Evansville, Indiana
  - Dermatology Clinical Trials Unit Washington University, St Louis, Missouri
  - Skin Specialists, PC, Omaha, Nebraska
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Dermatology Consulting Services, High Point, North Carolina
  - University Dermatology Consultants, Inc., Cincinnati, Ohio
  - Dermatology Research Associates Inc., Cincinnati, Ohio
  - Northwest Dermatology and Research Center, Portland, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - Paddington Testing Co., Inc., Philadelphia, Pennsylvania
  - Dermatology Research Association, Inc., Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - J&S Studies Inc., Bryan, Texas
  - Madison Skin & Research, Inc., Madison, Wisconsin